CLINICAL TRIAL: NCT06563544
Title: Flow Versus Volume-Controlled Ventilation in Intubated Obstructive and Asthmatic Patients
Brief Title: FCV Vs VCV in Obstructive and Asthmatic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maasstad Hospital (Other)
Responsible Party: Principal Investigator, Annemijn Jonkman, Dr. A.H. Jonkman, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ABR NL86078.078.24
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Pulmonary Disease; Mechanical Ventilation Pressure High; Asthma COPD
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Intervention Model Description: Physiological pilot study with a randomized crossover design comparing FCV and VCV
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FCV-VCV (Experimental): 90 minutes of FCV followed by 90 minutes of VCV
  Interventions: Device: FCV
- VCV-FCV (Experimental): 90 minutes of VCV followed by 90 minutes of FCV
  Interventions: Device: FCV

INTERVENTIONS:
Device: FCV — 90 minutes of FCV
  Other Names: Flow-controlled ventilation

SUMMARY:
The goal of this physiological pilot study with a randomized crossover design is to study the effect of Flow-controlled ventilation (FCV) on the minute volume compared to Volume-controlled ventilation (VCV) in intubated patients with an exacerbation of their asthma or COPD.

Our hypothesis is that FCV will results in a lower minute volume compared to VCV in this patient category.

Patients will be randomized between two ventilation sequences, namely 90 minutes of FCV followed by 90 minutes of VCV or vice versa.

DETAILED DESCRIPTION:
Rationale: Patients with an exacerbation of asthma or chronic obstructive pulmonary disease (COPD) requiring controlled mechanical ventilation (CMV) on the intensive care unit (ICU) have a mortality rate between 10 and 20%. This mortality rate is largely explained by major complications associated with mechanical ventilation e.g., pneumothorax, cardiovascular collapse and pneumonia. Complications are the result of dynamic hyperinflation that forms the cornerstone in the pathophysiology of both diseases. The diameter of the smaller airways decreases because of inflammation, bronchospasm, mucus (asthma) and the loss of elastic recoil by emphysema (COPD). This leads in particular to a high airway resistance during expiration and the residue of tidal volume in the lung when the next inspiration begins. The result is dynamic hyperinflation with a continuously increasing lung volume with high pressures, pneumothorax (barotrauma) and hemodynamic collapse as a result. During CMV (pressure- or volume controlled ventilation; PCV or VCV) only the inspiration is controlled while expiration is passive, possibly leading to airway collapse and further dynamic hyperinflation. Besides, both ventilation modes are accompanied by high flow rates leading to a further increase in airway resistance and ventilation pressures. Flow controlled ventilation (FCV) is a mechanical ventilation method that uses a relatively low and constant flow during both inspiration and expiration, thereby decreasing airway resistance and preventing airway collapse during expiration. Besides, FCV has shown to have a higher ventilation efficiency measured by a decrease in minute volume at stable arterial partial pressures of carbon dioxide (PaCO2). This makes FCV a very interesting ventilation mode in intubated patients with an exacerbation of asthma or COPD, possibly decreasing the amount of dynamic hyperinflation and complications in these patients. Although FCV is widely used for hypoxic respiratory failure on the ICU so far no studies have been performed in asthma or COPD patients.

We hypothesize that FCV in intubated patients with an exacerbation of asthma or COPD results in a lower minute volume (MV) and decreased end-inspiratory lung volume (EILV) as a measurement for dynamic hyperinflation compared to VCV.

Objectives: To study the effect of FCV on the MV and EILV compared to VCV.

Study design: Physiological pilot study with a randomized crossover design comparing FCV and VCV.

Study population: Patients with an asthma/COPD exacerbation ≥18 years old receiving CMV.

Intervention: Patients are mechanically ventilated with VCV at baseline. Upon inclusion the EIT-belt and an esophageal balloon are placed to assess the EILV and transpulmonary pressures respectively. Besides, patients are randomized between the sequence of ventilation mode, namely 90 minutes of VCV followed by 90 minutes of FCV or 90 minutes of FCV followed by 90 minutes of VCV. When VCV is switched to FCV the same mechanical ventilator settings are used as in the VCV mode. After half an hour on FCV the PEEP, drivingpressure and flow of FCV are optimized based on the highest compliance and lowest flow matching with a stable PaCO2. VCV is always set according to standard of care. Total time of measurements / study time is 180 minutes.

Main study parameters/endpoints: Primary endpoint is the difference in minute volume after 90 minutes on FCV compared to after 90 minutes of VCV. An important secondary endpoint is the difference in EILV after 30 minutes on FCV compared to after 30 minutes of VCV.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients are sedated and on CMV, therefore there will be no discomfort for the patient. FCV has been successfully applied during surgery and on the ICU and the patient will be monitored continuously so the clinical team can act directly in case of any adverse event. Lung volume is measured with EIT, a non-invasive, radiation-free monitoring tool. Transpulmonary pressures are measured with an esophageal balloon that is placed in a similar manor as a nasogastric feeding tube. Therefore, overall the risks of this study are limited.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Provided written informed consent;
* Undergoing controlled mechanical ventilation via an endotracheal tube;
* Reason for intubation being exacerbation of asthma or COPD;
* Intubated ≤72 hours

Exclusion Criteria:

* Severe sputum stasis or production requiring frequent bronchial suctioning (more than 5 times per nurse shift)
* Untreated pneumothorax (i.e. no pleural drainage)
* Hemodynamic instability defined as a mean arterial pressure below 60mmHg not responding to fluids and/or vasopressors or a noradrenalin dose >0.5mcrg/kg/min
* High (>15 mmHg) or instable (an increase in sedation or osmotherapy is required) intracranial pressure
* An inner tube diameter of 6mm or less
* Anticipating withdrawal of life support and/or shift to palliation as the goal of care
* Inability to perform adequate electrical impedance tomography (EIT) measurements with, e.g.:

  * Have a thorax circumference inappropriate for EIT-belt
  * Thoracic wounds, bandages or deformities preventing adequate fit of EIT-belt
  * Recent (<7 days) pulmonary surgery including pneumonectomy, lobectomy or lung transplantation
  * ICD device present (potential interference with proper functioning of the EIT device and ICD device)
  * Excessive subcutaneous emphysema
* Contra-indications for nasogastric tube or inability to perform adequate transpulmonary pressure measurements with, e.g.:

  * Recent esophageal surgery
  * Prior esophagectomy
  * Known presence of esophageal varices
  * Severe bleeding disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
MV | 90 minutes
  Minute Volume

SECONDARY OUTCOMES:
EILV | 90 minutes
  End-inspiratory lung volume
Vei | 90 minutes
  Volume end-inspiratory
MP | 90 minutes
  Mechanical Power (J/min)
Dissipated energy | 30 and 90 minutes
Airway pressures | 30 and 90 minutes
  (peak airway pressure, plateau pressure, mean airway pressure, PEEP, intrinsic PEEP, driving pressure
Transpulmonary pressures | 30 and 90 minutes
  (end-expiratory transpulmonary pressure, end-inspiratory transpulmonary pressure, transpulmonary driving pressure
RVDI | 30 and 90 minutes
  Regional ventilation delay index
GI | 30 and 90 minutes
  Global Inhomogeneity index
Gas exchange | 30 and 90 minutes
  Arterial blood gas values, ventilatory ratio
Hemodynamic parameters | 30 and 90 minutes
  Pulse rate and mean blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Diederik P Gommers, Prof. Dr., Study Director — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Maasstad Hospital, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed the researchers will deliver the study data to other researchers if asked for with good argumentation
Supporting Information: Study Protocol, SAP
Time Frame: After study completion
Access Criteria: Against good argumentation on request